CLINICAL TRIAL: NCT00669266
Title: Investigation of the Tumorigenesis of Adrenal Tumors and Evaluation of New Therapeutic Options - Untersuchungen Zur Tumorgenese Von Nebennierentumoren Und Evaluation Neuer Therapieoptionen
Brief Title: Adrenal Tumors - Pathogenesis and Therapy
Status: Recruiting | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Martin Fassnacht, Head of Endocrinology, University of Wuerzburg
Other Study IDs: Wue-Adrenal-Tumors-92/2002
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Adrenal Tumors; Adrenocortical Carcinoma; Cushing Syndrome; Conn Syndrome; Pheochromocytoma
MeSH Terms: conditions — Adrenal Gland Neoplasms; Adrenocortical Carcinoma; Cushing Syndrome; Hyperaldosteronism; Pheochromocytoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Germline DNA Tumor samples Serum Plasma Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tumor: Tumor material and corresponding biosamples from patients with adrenal tumors
- control group: Biomaterial from patients without adrenal tumor

SUMMARY:
The pathogenesis of adrenal tumors is still not fully elucidated and the treatment options for malignant tumors are poor. The current study investigates different aspects of the pathogenesis of adrenal tumors and evaluates different therapeutic options in patients with adrenocortical carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* adrenal tumor detected by imaging

Exclusion Criteria:

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with adrenal tumors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2002-09 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Principal Investigator — U of Wuerzburg
Locations (1):
- University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Result] Tamburello M, Altieri B, Sbiera I, Sigala S, Berruti A, Fassnacht M, Sbiera S. FGF/FGFR signaling in adrenocortical development and tumorigenesis: novel potential therapeutic targets in adrenocortical carcinoma. Endocrine. 2022 Sep;77(3):411-418. doi: 10.1007/s12020-022-03074-z. Epub 2022 May 18. PMID 35583844
- [Result] Sbiera I, Kircher S, Altieri B, Lenz K, Hantel C, Fassnacht M, Sbiera S, Kroiss M. Role of FGF Receptors and Their Pathways in Adrenocortical Tumors and Possible Therapeutic Implications. Front Endocrinol (Lausanne). 2021 Dec 9;12:795116. doi: 10.3389/fendo.2021.795116. eCollection 2021. PMID 34956100
- [Result] Weigand I, Ronchi CL, Vanselow JT, Bathon K, Lenz K, Herterich S, Schlosser A, Kroiss M, Fassnacht M, Calebiro D, Sbiera S. PKA Calpha subunit mutation triggers caspase-dependent RIIbeta subunit degradation via Ser114 phosphorylation. Sci Adv. 2021 Feb 19;7(8):eabd4176. doi: 10.1126/sciadv.abd4176. Print 2021 Feb. PMID 33608270
- [Result] Weigand I, Schreiner J, Rohrig F, Sun N, Landwehr LS, Urlaub H, Kendl S, Kiseljak-Vassiliades K, Wierman ME, Angeli JPF, Walch A, Sbiera S, Fassnacht M, Kroiss M. Active steroid hormone synthesis renders adrenocortical cells highly susceptible to type II ferroptosis induction. Cell Death Dis. 2020 Mar 17;11(3):192. doi: 10.1038/s41419-020-2385-4. PMID 32184394
- [Result] Ronchi CL, Di Dalmazi G, Faillot S, Sbiera S, Assie G, Weigand I, Calebiro D, Schwarzmayr T, Appenzeller S, Rubin B, Waldmann J, Scaroni C, Bartsch DK, Mantero F, Mannelli M, Kastelan D, Chiodini I, Bertherat J, Reincke M, Strom TM, Fassnacht M, Beuschlein F; European Network for the Study of Adrenocortical Tumors (ENSAT). Genetic Landscape of Sporadic Unilateral Adrenocortical Adenomas Without PRKACA p.Leu206Arg Mutation. J Clin Endocrinol Metab. 2016 Sep;101(9):3526-38. doi: 10.1210/jc.2016-1586. Epub 2016 Jul 7. PMID 27389594
- [Result] Beuschlein F, Fassnacht M, Assie G, Calebiro D, Stratakis CA, Osswald A, Ronchi CL, Wieland T, Sbiera S, Faucz FR, Schaak K, Schmittfull A, Schwarzmayr T, Barreau O, Vezzosi D, Rizk-Rabin M, Zabel U, Szarek E, Salpea P, Forlino A, Vetro A, Zuffardi O, Kisker C, Diener S, Meitinger T, Lohse MJ, Reincke M, Bertherat J, Strom TM, Allolio B. Constitutive activation of PKA catalytic subunit in adrenal Cushing's syndrome. N Engl J Med. 2014 Mar 13;370(11):1019-28. doi: 10.1056/NEJMoa1310359. Epub 2014 Feb 26. PMID 24571724